CLINICAL TRIAL: NCT02780973
Title: Influence of Gender Specific Differences of Saliva Composition on the Development of Dental Erosion - an In-situ Study
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Other Study IDs: Erosion-Gender; 7/10/15 (Other: Local Ethics Commission); 01681 (Other: UMG study center)
Record Dates: First submitted 2016-05-09; First posted 2016-05-24 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are obtained and retained for 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females: Female volunteers
  Interventions: Other: Wearing of an intraoral device with bovine tooth samples
- Males: Male volunteers
  Interventions: Other: Wearing of an intraoral device with bovine tooth samples

INTERVENTIONS:
Other: Wearing of an intraoral device with bovine tooth samples — Wearing of an intraoral device with bovine tooth samples

SUMMARY:
Healthy volunteers are observationally wearing an intraoral device with bovine tooth samples once for two hours. Afterwards, Calcium release from the bovine enamel and dentin samples is measured after extraoral erosion.

Total protein concentration within the formed salivary pellicles on the bovine samples is determined. Further Salivary parameters (unstimulated and stimulated saliva flow rate, pH, buffer capacity, albumin and total protein content as well as concentration of inorganic calcium, phosphate and fluoride) are being measured.

The aim of this study is to investigate whether gender differences in the salivary composition correlate with predisposition to erosion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy probands aged between 20 and 40 years who are able to give written consent

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Smoking
* Hyposalivation / xerostomia (unstimulated saliva < 0.3 mL/min, stimulated saliva < 0.7 mL/min)
* Intake of any medication (except contraceptives in women)
* Pregnant or lactating women
* Known allergies to substances used in the study
* Orthodontic treatment or malfunction which doesn't allow to wear an intraoral device

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Exploratory study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Calcium release from bovine enamel and dentin samples by extraoral erosion (nmol/Square Millimeter). | Immediately after the intraoral device has been worn once for two hours.

SECONDARY OUTCOMES:
Determination of unstimulated and stimulated saliva flow rate (mL/min). | Saliva samples are collected for 5 min each on two visits.
Determination of saliva pH. | Saliva samples are collected for 5 min each on two visits.
Determination of salivary buffer capacity. | Saliva samples are collected for 5 min each on two visits.
Determination of albumin (mg/L) in saliva. | Saliva samples are collected for 5 min each on two visits.
Determination of total protein content (mg/L) in saliva. | Saliva samples are collected for 5 min each on two visits.
Determination of inorganic calcium (mmol/l), phosphate (mmol/L) and fluoride (µmol/L) in saliva. | Saliva samples are collected for 5 min each on two visits.
Determination of total protein concentration in the formed salivary pellicles (ng/Square Millimeter). | Immediately after the intraoral device has been worn once for two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prodan A, Brand HS, Ligtenberg AJ, Imangaliyev S, Tsivtsivadze E, van der Weijden F, Crielaard W, Keijser BJ, Veerman EC. Interindividual variation, correlations, and sex-related differences in the salivary biochemistry of young healthy adults. Eur J Oral Sci. 2015 Jun;123(3):149-57. doi: 10.1111/eos.12182. Epub 2015 Mar 23. PMID 25809904
- [Background] Carpenter G, Cotroneo E, Moazzez R, Rojas-Serrano M, Donaldson N, Austin R, Zaidel L, Bartlett D, Proctor G. Composition of enamel pellicle from dental erosion patients. Caries Res. 2014;48(5):361-7. doi: 10.1159/000356973. Epub 2014 Mar 6. PMID 24603346
- [Background] Moazzez R, Bartlett D. Intrinsic causes of erosion. Monogr Oral Sci. 2014;25:180-96. doi: 10.1159/000360369. Epub 2014 Jun 26. PMID 24993266
- [Background] Wiegand A, Bliggenstorfer S, Magalhaes AC, Sener B, Attin T. Impact of the in situ formed salivary pellicle on enamel and dentine erosion induced by different acids. Acta Odontol Scand. 2008 Aug;66(4):225-30. doi: 10.1080/00016350802183401. PMID 18607835
- [Background] Wiegand A, Meier W, Sutter E, Magalhaes AC, Becker K, Roos M, Attin T. Protective effect of different tetrafluorides on erosion of pellicle-free and pellicle-covered enamel and dentine. Caries Res. 2008;42(4):247-54. doi: 10.1159/000135669. Epub 2008 Jun 4. PMID 18523383
- [Background] Zwier N, Huysmans MC, Jager DH, Ruben J, Bronkhorst EM, Truin GJ. Saliva parameters and erosive wear in adolescents. Caries Res. 2013;47(6):548-52. doi: 10.1159/000350361. Epub 2013 Jun 15. PMID 23774653
- [Background] Kanzow P, Wegehaupt FJ, Attin T, Wiegand A. Etiology and pathogenesis of dental erosion. Quintessence Int. 2016 Apr;47(4):275-8. doi: 10.3290/j.qi.a35625. PMID 27022647
- [Result] Wiegand A, Rosemann A, Hoch M, Barke S, Dakna M, Kanzow P. Erosion-Protective Capacity of the Salivary Pellicle of Female and Male Subjects Is Not Different. Caries Res. 2019;53(6):636-642. doi: 10.1159/000500046. Epub 2019 Jun 4. PMID 31163440